CLINICAL TRIAL: NCT02401646
Title: Clinical Trials for the Effects of Polygoni Multiflori Radix Complex Extract on Memory Improvement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Memory_2015
Record Dates: First submitted 2015-02-25; First posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Memory, Short-Term

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polygoni Multiflori Radix complex (Experimental): Participants randomized to the experimental group will take one capsule of Polygoni Multiflori Radix complex extract (250mg) twice a day, 30 minutes after breakfast and dinner for 4 weeks.
  Interventions: Dietary Supplement: Polygoni Multiflori Radix complex extract
- Starch (Placebo Comparator): Participants randomized to the placebo group will take one capsule of placebo(250mg) twice a day, 30 minutes after breakfast and dinner for 4 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Polygoni Multiflori Radix complex extract — Intervention is manufactured by Chun-Ho food
  Arms: Polygoni Multiflori Radix complex
Dietary Supplement: Placebo — The placebo is filled with starch, so does not contain the active ingredient.
  Arms: Starch

SUMMARY:
The aim of this study is to identify the effect of Polygoni Multiflori Radix complex extract on memory improvement using Rey-Kim scale for healthy people.

ELIGIBILITY:
Inclusion Criteria:

* A person who is more than 50 years and lesser than 70 years of age
* A person who's MQ(Memory Quotient) score is within more than 70 and lesser than 120

Exclusion Criteria:

* The patient who has past history related to memory
* The patient who has Diabetes Mellitus
* The person whose fasting blood sugar is more than 126mg/dL
* The patients who has uncontrolled hypertension
* The patient who has liver disorders
* The patient whose AST(aspartate aminotransferase) or ALT(alanine aminotransferase) level is more than 60 IU/L(international units per liter)
* The patients who has heart disorders (Angina pectoris, Myocardial infarction)
* The patient who has past history related to excision of G-I tract excluding cecum
* The patient who took drug or heal functional food within 4 weeks before screening
* The patient who took decoction of herb within 4 weeks before screening
* The patient who can't write or communicate
* pregnant woman

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on Memory Quotient score at 2 weeks and 4 weeks | baseline, at 2 weeks after taking experimental or placebo dietary supplement, at 4 weeks after taking supplement

SECONDARY OUTCOMES:
Change from baseline in Memory registration at 2 weeks and 4 weeks | baseline, at 2 weeks after taking experimental or placebo dietary supplement, at 4 weeks after taking supplement
  Rey-Kim scale is a tool to assess the short-term memory. It is composed of AVLT and CFT.
  # AVLT After tester speaks each 15 word, subjects are asked to tell all words immediately as memory serves. This process is repeated 5 times (Each process is called AVLT process 1-5 according to priority). After 20 minutes interval, subjects are also asked to tell all words they can remember (AVLT process 6). Right after that, subjects should select the words they heard among 35 words (AVLT process 7).
  Memory registration is calculated by converting score difference into a percentage between AVLT process 1 and 5 mentioned above.
Change from baseline in Memory retention at 2 weeks and 4 weeks | baseline, at 2 weeks after taking experimental or placebo dietary supplement, at 4 weeks after taking supplement
  # AVLT After tester speaks each 15 word, subjects are asked to tell all words immediately as memory serves. This process is repeated 5 times (Each process is called AVLT process 1-5 according to priority). After 20 minutes interval, subjects are also asked to tell all words they can remember (AVLT process 6). Right after that, subjects should select the words they heard among 35 words (AVLT process 7).
  Memory retention is calculated by converting score difference into a percentage between AVLT process 5 and 6 mentioned above.
Change from baseline in Retrieval efficiency at 2 weeks and 4 weeks | baseline, at 2 weeks after taking experimental or placebo dietary supplement, at 4 weeks after taking supplement
  # AVLT After tester speaks each 15 word, subjects are asked to tell all words immediately as memory serves. This process is repeated 5 times (Each process is called AVLT process 1-5 according to priority). After 20 minutes interval, subjects are also asked to tell all words they can remember (AVLT process 6). Right after that, subjects should select the words they heard among 35 words (AVLT process 7).
  Retrieval efficiency is calculated by converting score difference into a percentage between AVLT process 6 and 7 mentioned above.
Change from baseline in Copy-recall difference index at 2 weeks and 4 weeks | baseline, at 2 weeks after taking experimental or placebo dietary supplement, at 4 weeks after taking supplement
  Rey-Kim scale is a tool to assess the short-term memory. It is composed of AVLT and CFT.
  # CFT After tester shows subjects very complicated figure, subjects are asked to copy it (CFT process 1). Right after that, subjects should draw the figure as memory serves (CFT process 2). After 20 minutes interval, subjects are also asked to select the part of figure they copy among various figures (CFT process 3).
  Copy-recall difference index is calculated by converting score difference into a percentage between CFT process 1 and 2 mentioned above.

CONTACTS AND LOCATIONS:
Overall Officials: In Lee, Doctor, Study Chair — Pusan National University Korean Medicine Hospital; Hye-lim Park, Master, Principal Investigator — Pusan National University Korean Medicine Hospital; Eunhye Jeong, bachelor, Principal Investigator — National Clinical Research Center for Korean Medicine Pusan National University Korean Medicine Hospital; Hana Lee, bachelor, Principal Investigator — National Clinical Research Center for Korean Medicine Pusan National University Korean Medicine Hospital
Locations (1):
- Pusan National University Korean Medicine Hospital, Yangsan, Gyeongsangnam-do, South Korea